CLINICAL TRIAL: NCT02443753
Title: A Pilot Safety and Tolerability Study of the Use of the EndoBarrier® SANS™ in Over-weight or Obese Type 2 Diabetic Subjects
Brief Title: EndoBarrier® SANS™ in Over-weight or Obese Type 2 Diabetic Subjects
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Morphic Medical Inc. (Industry)
Collaborators: University of Malaya (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15-1
Record Dates: First submitted 2015-05-11; First posted 2015-05-14 (Estimated); Last update posted 2016-02-10 (Estimated); Status verified 2016-02

CONDITIONS: Obesity; Type 2 Diabetes
MeSH Terms: conditions — Obesity; Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Device (Experimental): Subjects who receive the device
  Interventions: Device: EndoBarrier SANS

INTERVENTIONS:
Device: EndoBarrier SANS — Eligible subjects will be implanted with the EndoBarrier® SANS™ Device for a period of 3 months. The GI Dynamics' EndoBarrier® SANS™ is an endoscopically positioned device that represents an alternative to the use of gastric bypass operative techniques as a means of re-routing food and altering the gut-hormone axis. The EndoBarrier® SANS™ provides an alternate passage of chime through the duodenum and proximal sixty centimeters of jejunum replicating in part the bypass of bariatric surgery.

SUMMARY:
This study will evaluate the safety and efficacy of the EndoBarrier® SANS™ in overweight and obese subjects with type 2 diabetes. The barbless second generation device is being developed as a means to reduce the incidence of adverse events associated with the barbs of the predicate device while maintaining a similar efficacy profile as measured by changes in weight and diabetic endpoints (HbA1c, blood glucose, insulin, etc.). This first use in human will primarily evaluate preliminary safety, tolerability and efficacy of the new design. Because of the new design and its first study in human subjects, only a 3 month implant duration will be evaluated in this study.

DETAILED DESCRIPTION:
The GI Dynamics' EndoBarrier® SANS™ is an endoscopically positioned device that represents an alternative to the use of gastric bypass operative techniques as a means of re-routing food and altering the gut-hormone axis. The EndoBarrier® SANS™ provides an alternate passage of chime through the duodenum and proximal sixty centimeters of jejunum replicating in part the bypass of bariatric surgery.

This study will be conducted at a single clinical site in Malaysia. Approximately 16 subjects will be enrolled in two cohorts of 8 subjects. The two cohorts will be implanted one week apart with the implantation of the second cohort triggered by the absence of major technical or clinical issues (i.e. safety, tolerability) observed in the first cohort in the first seven days.

ELIGIBILITY:
Inclusion Criteria:

* Age > 21 years and < 65 years - male or female
* Overweight or obese individuals (BMI ≥ 27 kg/m2 and ≤ 40 kg/m2)
* Diagnosed with Type 2 diabetes and being treated by diet or oral agents (metformin, SU, DPP-4i, or TZD)
* Glycemic state: HbA1c at screening 7.0-10.0%.
* History of failure with non-surgical weight loss methods
* Subjects willing to comply with study requirements
* Subjects who have signed an informed consent form

Exclusion Criteria:

Diabetic subjects requiring injectable treatments (insulin, GLP-1R agonists)

* Subjects requiring anticoagulation therapy
* Subjects with iron deficiency and iron deficiency anemia
* Condition of the gastrointestinal tract, such as ulcers or inflammatory bowel disease
* Treatment represents an unreasonable risk to the subject
* Known history of acute or chronic pancreatitis
* Known history of organ failure (i.e. renal insufficiency, heart failure, fibrotic / cirrhotic liver disease, or pulmonary disease)
* Symptomatic coronary artery disease or pulmonary dysfunction
* Subjects with known symptomatic biliary disease
* Known infection at the time of implant
* Severe coagulopathy, upper gastro-intestinal bleeding conditions such as esophageal or gastric varices, congenital or acquired intestinal telangiectasia
* Congenital or acquired anomalies of the GI tract such as atresias or stenoses
* Pregnant or has the intention of becoming pregnant in the next 6 months
* Unresolved alcohol or drug addiction
* HIV positive subjects
* Subjects with hepatitis B or C
* Currently taking the following medications within 30 days of implant:

systemic corticosteroids, drugs known to affect GI motility, prescription or over the counter weight loss medications such as Sibutramine hydrochloride monohydrate and Orlistat

* Allergy or hypersensitivity to ceftriaxone, cephalosporins, penicillin, and all equivalent antibiotics
* Any characteristics which, in the opinion of the investigator, makes the subject a poor candidate for device placement in this clinical trial
* Previous GI surgery that could affect the ability to place the liner or the function of the implant.
* Subjects unable to discontinue NSAIDs (non-steroidal anti-inflammatory drugs) during the implant period
* H. pylori positive subjects (Note: patients may be enrolled if they had a prior history and were successfully treated).
* Family or subject history of a known diagnosis or pre-existing symptoms of systemic lupus erythematosus, scleroderma or other autoimmune connective tissue disorder
* Unable to tolerate proton pump inhibitors
* Participating in another ongoing investigational clinical trial that is ongoing or within 3 months of the implant date
* Positive stool guaiac at time of screening

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2015-05; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Safety and Tolerability will be evaluated as the incidence of AEs and SAEs/UADEs. | 3 months
  Safety will be evaluated as the incidence of AEs and SAEs/UADEs.

SECONDARY OUTCOMES:
Efficacy as measured by Change in Body weight | 3 months
  Change in Body weight
Efficacy as measured by Percent excess weight loss | 3 months
  Percent excess weight loss
Efficacy as measured by Change in HbA1c (%) | 3 months
  Change in HbA1c (%)

CONTACTS AND LOCATIONS:
Overall Officials: Eng Hong Pok, MD, Principal Investigator — University of Malaya; Wah Kheong Chan, MD, Principal Investigator — University of Malaya
Locations (1):
- Universiti Malaya Medical Centre, Jalan universiti, Kuala Lumpur, Malaysia